CLINICAL TRIAL: NCT06814132
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MK-5684 in Male Participants With Severe Renal Impairment and With End-stage Renal Disease
Brief Title: A Study to Evaluate the Effect of MK-5684 in Male Participants With Severe Renal Impairment (RI) and With End-stage Renal Disease (ESRD) (MK-5684-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5684-010; MK-5684-010 (Other: MSD); CA43216 (Other: Celerion)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Kidney Failure, Chronic; End-Stage Kidney Disease; Renal Failure, Chronic; Renal Failure, End-Stage; Healthy Participants
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Prednisone; fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Severe Renal Impairment (RI) (Experimental): Participants will receive a single oral dose of MK-5684 under fasting conditions (on an empty stomach after a 10-hour overnight fast) on Day 1 and a single dose of Hormone replacement therapy (HRT) (prednisone and fludrocortisone) administered approximately 4.5 hours after MK-5684 dosing under fed conditions (eating a normal meal).
  Interventions: Drug: MK-5684; Drug: Prednisone; Drug: Fludrocortisone acetate
- Group 2: End-stage renal disease (ESRD) (Experimental): Participants will receive a single oral dose of MK-5684 under fasting conditions (on an empty stomach after a 10-hour overnight fast) in Period 1 and Period 2. In Period 1, participants will receive a single oral dose of MK-5684 approximately 30 minutes prior to their normally scheduled hemodialysis (HD), followed by HRT under fed conditions (eating a normal meal) 4.5 hours after MK-5684 dosing. In Period 2, participants will receive a single oral dose of MK-5684 immediately followed by completion of their normally scheduled HD, and by HRT under fed conditions (eating a normal meal) 4.5 hours after MK-5684 dosing.
  Interventions: Drug: MK-5684; Drug: Prednisone; Drug: Fludrocortisone acetate
- Group 3: Healthy Participants (Experimental): Participants will receive a single oral dose of MK-5684 under fasting conditions (on an empty stomach after a 10-hour overnight fast) on Day 1 and a single dose of Hormone replacement therapy (HRT) (prednisone and fludrocortisone) administered approximately 4.5 hours after MK-5684 dosing under fed conditions (eating a normal meal).
  Interventions: Drug: MK-5684; Drug: Prednisone; Drug: Fludrocortisone acetate

INTERVENTIONS:
Drug: MK-5684 — Oral tablet
Drug: Prednisone — Oral tablet
  Other Names: HRT
Drug: Fludrocortisone acetate — Oral tablet
  Other Names: HRT

SUMMARY:
The goal of the study is to learn what happens to levels of MK-5684 in people with severe renal impairment and end-stage renal disease versus a healthy person's body over time. Researchers will compare what happens to MK-5684 after hemodialysis in people with severe renal impairment and end-stage renal disease versus healthy people.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

All Participants

* Is a continuous non-smoker or moderate smoker (≤ 10 cigarettes per day or equivalent) for at least 3 months prior to the first dosing
* Has a body mass index (BMI) ≥ 18.0 and ≤ 42.0 kg/m^2 at the screening visit

Participants with severe renal impairment (RI) (Group 1):

* Has severely impaired renal function as determined by estimated glomerular filtration rate (eGFR) using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation

Participants with end-stage renal disease (ESRD) (Group 2):

* Has ESRD maintained on stable outpatient regimen of intermittent high-flux hemodialysis (HD) (at least 3 times per week) for a minimum of 3 hours per dialysis session, using a complication free well-maintained arteriovenous fistula or arteriovenous graft, for at least 3 months prior to first dosing and is expected and planning to continue HD during the study and at least up to the follow-up visit

Healthy Control Participants (Group 3):

* Has normal renal function

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

All Participants:

* Has a history or presence of any of the following: Adrenal insufficiency; Hepatic impairment; Clinically significant hypotension; cardiac arrhythmia; cardiac conduction abnormalities or recurrent unexplained syncopal events; Second- or third-degree atrioventricular (AV) heart block (except in participants with a functional artificial pacemaker); Clinically significant sick sinus syndrome; Any systemic fungal infection; Hypothyroidism; Chronic infection
* Has a first-degree relative with multiple unexplained syncopal events, unexplained cardiac arrest, or sudden cardiac death, or has a known family history of an inherited arrhythmia syndrome (including Brugada syndrome)
* Has a history of cancer (malignancy)
* Is positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)

Participants with Severe RI (Group 1):

* Has a history or presence of renal artery stenosis
* Has had a renal transplant
* Has ESRD requiring HD

Participants with ESRD (Group 2):

* Has required frequent emergent HD (≥ 3) within a year prior to the first dosing
* Has a history or presence of renal artery stenosis.
* Has had a functioning renal transplant within the past 2 years

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve from 0 to Infinity (AUC0-inf) After a Single Dose of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the AUC0-inf of MK-5684 in plasma.
Area Under the Concentration Versus Time Curve From 0 to the Time of the Last Quantifiable Sample (AUC0-last) of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the AUC0-last of MK-5684 in plasma.
Area Under the Concentration Versus Time Curve From 0 to 24 Hours After Dosing (AUC0-24) of MK-5684 | At protocol specific time points pre-dose and up to 24 hours post-dose
  Blood samples will be collected to determine the AUC0-24 of MK-5684 in plasma.
Maximum Observed Drug Concentration (Cmax) After the Administration of a Given Dose of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the Cmax of MK-5684 in plasma.
Time to Maximum Observed Plasma Drug Concentration (Tmax) of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the Tmax of MK-5684 in plasma.
Apparent Terminal Half-Life (t½) of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the t1/2 of MK-5684 in plasma.
Apparent Clearance (CL/F) of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the CL/F of MK-5684 in plasma.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-5684 | At protocol specific time points pre-dose and up to 72 hours post-dose
  Blood samples will be collected to determine the Vz/F of MK-5684 in plasma.

SECONDARY OUTCOMES:
Number of Participants who Experience an Adverse Event (AE) | Up to ~21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to ~7 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Dialysis Clearance (CLD) of MK5684 Based on Plasma | At protocol specific time points pre-dose and up to 4.5 hours post-dose
  Dialysate will be collected to determine the CLD of MK-5684 in plasma.
Concentration of Dialysate (CD) of MK-5684 Samples | At protocol specific time points pre-dose and up to 4.5 hours post-dose
  Dialysate will be collected to determine the CD of MK-5684 in plasma.
Amount of drug (AD) of MK-5684 recovered from each dialysate collection | At protocol specific time points pre-dose and up to 4.5 hours post-dose
  Dialysate will be collected to determine the AD of MK-5684 in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida
  - Research by Design ( Site 0001), Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/